CLINICAL TRIAL: NCT06946199
Title: An Open-label Study Evaluating the Safety and Preliminary Clinical Activity of Cizutamig in Patients With Refractory Seropositive Rheumatoid Arthritis
Brief Title: An Open-label Study of Cizutamig in Refractory Seropositive Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Qiubai Li, Director, Head of Department of Rheumatology and Immunology, Principal Investigator, Professor, Wuhan Union Hospital, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT250171
Record Dates: First submitted 2025-04-10; First posted 2025-04-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: cizutamig; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cizutamig (Experimental)
  Interventions: Drug: Cizutamig; Biological: Cizutamig

INTERVENTIONS:
Drug: Cizutamig — Cizutamig will be administered per the dose escalation cohort
Biological: Cizutamig — Cizutamig will be administered per the dose escalation cohort

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of BCMAxCD3 T-cell engager (cizutamig) in patients with refractory seropositive RA.

DETAILED DESCRIPTION:
B cells mature into plasmablasts and plasma cells that are prolific antibody producers and the predominant source of pathogenic autoantibodies, a hallmark of RA. Autoantibodies contribute to the pathogenesis of RA in several ways, including formation of immune complexes, activation of complement and downstream cell lysis. Clinical trials of cizutamig (BCMAxCD3 T-cell engager) demonstrated safety and efficacy in RRMM. Cizutamig offers a promising mechanism of action for refractory seropositive RA. This study aims to assess the safety, tolerability, PK, pharmacodynamics, immunogenicity, and preliminary clinical activity of cizutamig administered in patients with refractory seropositive RA. Patients will be invited to participate in the study, to receive cizutamig and monitored after dosing with cizutamig through Week 52.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old at the time of signing the informed consent form
2. Diagnosis of adult-onset RA as defined by the 2010 ACR/EULAR classification criteria
3. Moderately to severely active RA.
4. Positive test results for RF and/or ACPA at Screening.

Inadequate treatment response defined as either lack of clinical benefit or intolerability to treatment with tsDMARD and/or bDMARD Exclusion Criteria:

1. Inadequate clinical laboratory parameters at Screening
2. Patients with active infection
3. Receipt of live vaccine within 4 weeks prior to Screening
4. Presence of any concomitant autoimmune disease
5. History of progressive multifocal leukoencephalopathy
6. History of primary immunodeficiency or a hereditary deficiency of the complement system
7. Central nervous system disease
8. Presence of 1 or more significant concurrent medical conditions per investigator judgment
9. Have a diagnosis or history of malignant disease within 5 years
10. Serious mental illness, alcohol or drug abuse, dementia, or any other condition that would impair the patient's ability to receive the planned treatment or to understand informed consent at the study site as determined by local practice

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events through end of study | Baseline to Month 12
  Incidence and severity of TEAEs through end of study.
Changes from baseline in vital signs through end of study: body temperature | Baseline to Month 12
Changes from baseline in vital signs through end of study: heart rate | Baseline to Month 12
Changes from baseline in vital signs through end of study: respiratory rate | Baseline to Month 12
Changes from baseline in vital signs through end of study: blood pressure | Baseline to Month 12
Changes from baseline in vital signs through end of study: pulse oximetry | Baseline to Month 12
Changes from baseline in ECG parameters through end of study: PR interval | Baseline to Month12
Changes from baseline in ECG parameters through end of study: QRS interval | Baseline to Month 12
Changes from baseline in ECG parameters through end of study: QTcF interval | Baseline to Month 12
Changes from baseline in safety laboratory assessments through end of study: serum chemistry | Baseline to Month 12
Changes from baseline in safety laboratory assessments through end of study: hematology | Baseline to Month 12

SECONDARY OUTCOMES:
Pharmacokinetic (PK) for Cizutamig: Cmax | Baseline to Month 12
PK parameters for Cizutamig: time of maximum concentration | Baseline to Month 12
PK parameters for Cizutamig: area under the concentration-time curve | Baseline to Month 12
PK parameters for Cizutamig: clearance | Baseline to Month 12
PK parameters for Cizutamig: volume of distribution | Baseline to Month 12
PK parameters for Cizutamig: half-life | Baseline to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Qiubai Li, Professor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No